CLINICAL TRIAL: NCT02184507
Title: Effect of Insulin Resistance Reducing Agents Pre and Post CABG on Post-operative Metabolic Status and Oxidative Stress
Acronym: ECIRRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mohammad Hassan Eftekhari (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Mohammad Hassan Eftekhari, Professor. PhD, Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91-6447
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Coronary Artery Disease
Keywords: insulin resistance; blood glucose; CABG; oxidative stress
MeSH Terms: conditions — Coronary Artery Disease; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Supplement pre CABG (Experimental): Consumption of the supplement 7 days before surgery and placebo 30 days post surgery
  Interventions: Dietary Supplement: Supplement pre CABG
- Supplement post CABG (Experimental): Consumption of placebo 7 days before surgery and supplement 30 days post surgery
  Interventions: Dietary Supplement: Supplement post CABG
- Supplement pre and post CABG (Experimental): Consumption of the supplement 7 days before and 30 days post surgery
  Interventions: Dietary Supplement: Supplement pre and post CABG
- Placebo (Placebo Comparator): Consumption of placebo 7 days before and 30 days post surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement pre CABG — One sachet of the supplement was consumed daily for 7 days before surgery.
  Arms: Supplement pre CABG
Dietary Supplement: Supplement post CABG — One sachet of the supplement was consumed daily for 30 days after surgery
  Arms: Supplement post CABG
Dietary Supplement: Supplement pre and post CABG — One sachet of the supplement was consumed daily for 7 days before surgery and 30 days after CABG
  Arms: Supplement pre and post CABG
Drug: Placebo — One sachet of placebo was consumed daily for 7 days before surgery and 30 days after CABG
  Arms: Placebo

SUMMARY:
The present study aimed to evaluate the effect of a combination of insulin resistance reducing agents pre and post coronary artery bypass grafting surgery on post-operative blood glucose and oxidative stress regulation.

DETAILED DESCRIPTION:
The present study aimed to evaluate the effect of a combination of insulin resistance reducing agents pre and post coronary artery bypass grafting surgery on post-operative blood glucose and oxidative stress regulation. The sample size was estimated to be 92 (23 in each group). The participants of the study were selected from the non-diabetic patients scheduled for CABG. The patients were allocated to four groups using balanced block randomization method:

1. Consumption of the supplement (a 20 gram pack of the supplement daily) 7 days before surgery and placebo (a pack of starch) 30 days post surgery
2. Consumption of placebo 7 days before surgery and supplement 30 days post surgery
3. Consumption of the supplement 7 days before and 30 days post surgery
4. Consumption of placebo 7 days before and 30 days post surgery One week before, before the onset of the surgery, after the surgery, 1 week after and 4 weeks after the operation, blood samples were taken and the levels of hemoglobin A1C, glucose, insulin and malondialdehyde were measured. Also, body composition indices were assessed in four times: one week before the surgery, before the onset of the surgery, 1 week after and 4 weeks after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Mean age of 30-70 years old, Having Coronary Artery Disease
* Undergoing coronary artery bypass grafting surgery

Exclusion Criteria:

* Positive history of diabetes mellitus, metabolic, hematological, and immune disorders, renal problem, and cerebrovascular accident
* Taking antioxidant supplements
* Cases for emergency operations
* Ejection Fraction < 30%

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-06; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Serum glucose | 37days
  It was measured in 5 steps:
  1 week before the operation, Just before the operation, After operation, 1 week post operation, 30 days post operation
serum insulin | 37 days
  It was measured in 5 steps:
  1 week before the operation, Just before the operation, After operation, 1 week post operation, 30 days post operation
Hemoglobin A1C | 37 days
  It was measured in 4 steps:
  1 week before the operation, Just before the operation, 1 week post operation, 30 days post operation
Insulin Resistance | 37 days
  Calculated by HOMA calculation equation
  It was calculated in 5 steps:
  1 week before the operation, Just before the operation, After operation, 1 week post operation, 30 days post operation

SECONDARY OUTCOMES:
Body Composition changes | 37 days
  It was measured in 4 steps:
  1 week before the operation, Just before the operation, 1 week post operation, 30 days post operation
malondialdehyde | 37 days
  It was measured in 5 steps:
  1 week before the operation, Just before the operation, After operation, 1 week post operation, 30 days post operation

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hassan Eftekhari, professor, Study Director — Shiraz University of Medical Sciences